CLINICAL TRIAL: NCT04105530
Title: Transcranial Direct Current Stimulation of the Temporal Cortex in Survivors of Childhood Acute Lymphoblastic Leukemia (ALL)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: ALLSUP; NCI-2019-07041 (Registry Identifier: NCI)
Record Dates: First submitted 2019-06-25; First posted 2019-09-26 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Acute Lymphoblastic Leukemia; Transcranial Direct Current Stimulation; Executive Dysfunction
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: Enrollment is on hold per institutional COVID-19 guidelines
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Transcranial direct current stimulation (tDCS) on day 1 (Active Comparator): One stimulation will be conducted using Anodal treatment.
  The Direct Current Anodal Stimulation will be applied for 20 minutes for each stimulation period. Brief neurocognitive testing will be conducted during each stimulation session.
  Interventions: Device: Anodal tDCS treatment; Other: NIH Toolbox List Sorting Working Memory Test; Other: NIH Toolbox Flanker Inhibitory Control and Attention Test; Other: Grooved Peg Board Test; Other: Buschke Selective Reminding Test
- Transcranial direct current stimulation (tDCS) on day 2 (Active Comparator): A final stimulation will be conducted using Cathodal stimulation. Direct Current Cathodal Stimulation will be applied for 20 minutes for each stimulation period. Brief neurocognitive testing will be conducted during each stimulation session.
  Interventions: Device: Cathodal tDCS treatment; Other: NIH Toolbox List Sorting Working Memory Test; Other: NIH Toolbox Flanker Inhibitory Control and Attention Test; Other: Grooved Peg Board Test; Other: Buschke Selective Reminding Test
- Sham treatment (Placebo Comparator): The sham procedure provides the same small current during ramp up to imitate the intervention, but the current is discontinued after ramping up and no intervention is provided. Sham will be applied for 20 minutes.Stimulation will start 5 minutes before testing and continue throughout completing the NIH Toolbox Cognitive Battery at each trial:"
  Interventions: Device: Sham treatment; Other: NIH Toolbox List Sorting Working Memory Test; Other: NIH Toolbox Flanker Inhibitory Control and Attention Test; Other: Grooved Peg Board Test; Other: Buschke Selective Reminding Test

INTERVENTIONS:
Device: Anodal tDCS treatment — The Anodal intervention excites neuronal activity. For condition one, the anode will be attached to the left frontal region (Fp1) and the cathode will be attached to the right neck. The intervention involves a direct current of 1 mA applied for 20 minutes.
  Arms: Transcranial direct current stimulation (tDCS) on day 1
Device: Cathodal tDCS treatment — The Cathodal intervention inhibits or reduces neuronal activity. We propose that the use of the cathodal tDCS to the superior temporal gyrus in survivors of childhood ALL may facilitate the inhibition of over connected motor-sensory and auditory neural networks. For condition two, the cathode will be attached to the left temporal region (T3) and the anode will be attached to the right neck. The intervention involves a direct current of 1 mA applied for 20 minutes.
  Arms: Transcranial direct current stimulation (tDCS) on day 2
Device: Sham treatment — The sham procedure provides the same small current during ramp up to imitate the intervention, but the current is discontinued after ramping up and no intervention is provided. Sham will be applied for 20 minutes. Stimulation will start 5 minutes before testing and continue throughout completing the NIH Toolbox Cognitive Battery at each trial.
  Arms: Sham treatment
Other: NIH Toolbox List Sorting Working Memory Test — List Sorting is using information processing and storage. Performance tends to peak in early adulthood and then decline across the life span. This task assesses working memory and requires the participant to sequence different visually- and orally-presented stimuli. The list scoring task takes approximately 7 minutes to administer. List Sorting is scored by summing the total number of items correctly recalled and sequenced on Lists-1 and -2, which can range from 0-26.
Other: NIH Toolbox Flanker Inhibitory Control and Attention Test — The Flanker tests inhibitory control and attention and the capacity for new learning and information processing novel situations. This performance also reaches a peak in early adulthood and tends to decline across the life span. A total of 40 trials require 4 minutes. Scoring is based on both accuracy and reaction time, which will we evaluate individually as well as in combination. The raw scores are converted to a scale score with a mean of 100 and SD of 15. Higher scores indicate higher executive function.
Other: Grooved Peg Board Test — The Grooved Peg Board test measures visual-motor coordination and motor speed. Additionally, it is cognitively challenging and has been associated with attention, perceptual speed and non-verbal reasoning. Performance is better in the dominant/preferred hand and tends to improve in childhood and decline with advancing age. The test consists of placing metal pegs with ridges along onside in matching slots as quickly as possible. The score is the time in seconds required to compete the array with each hand. Longer times reflect worse performance. Times are compared to normative data that is organized by ethnicity, age, gender and education. The test takes approximately 5 minutes to complete.
Other: Buschke Selective Reminding Test — This selective reminding task purports to distinguish verbal memory into short-term and long-term components. Scores are organized by short- and long-term storage and retrieval with normative scores organized by age and gender. The task requires participants to remember a list of orally-presented words and recall them with selective reminders of the words that they didn't recall. The test will last 5-10 minutes and is available in four different versions, thus reducing rehearsal effects.

SUMMARY:
Brief Overview: Children and adolescents diagnosed with cancer will experience problems with learning, memory and attention during and after completing their cancer therapy. There are many factors that contribute to this problem, but investigators have recently identified that chemotherapy agents used in treating Acute Lymphoblastic Leukemia (ALL) may disrupt normal brain development.

A novel device has been developed that may help correct this disruption. Direct Current Stimulation (DCS) uses a very low level of constant electrical current to stimulate specific parts of the brain. It has been used in patients with stroke to great benefit. Our study at St. Jude Children's Research Hospital is designed to see if this technique will benefit survivors of childhood cancer. Specifically, investigators wish to see if stimulating one part of the brain gives a greater benefit than stimulating another part of the brain.

Primary Objective

Evaluate the feasibility of conducting repeated on-site Transcranial Direct Current Stimulation (tDCS) in children who are long-term survivors of

Secondary Objectives

* To estimate the potential efficacy for powering a future larger study using tDCS to improve cognitive performance in children by suppressing over connected neural hubs in long-term survivors of childhood ALL.
* To compare the performance of anodal stimulation of the frontal lobe to cathodal suppression of the superior temporal lobe on cognitive performance.

DETAILED DESCRIPTION:
Participants will be randomly assigned to one of three intervention arms. Two brief stimulation periods will be conducted on day one. One brief stimulation will be scheduled in the morning and a second brief stimulation will be scheduled in the afternoon. A final stimulation will be conducted on day two. Direct Current Stimulation will be applied for 20 minutes for each stimulation period. Brief neurocognitive testing will be conducted during each stimulation session.

ELIGIBILITY:
Inclusion Criteria:

* ALL survivors who received chemotherapy-only treatment and are enrolled in SJLIFE.
* 8-17 years old.
* History of executive function, processing speed and/or memory impairment documented as a score < 10th percentile of the age adjusted Z-score.
* Participants able to speak and understand the English language.

Exclusion Criteria:

* Survivors who received cranial radiation.
* Survivors with a Full-Scale IQ < 70.
* Pregnant, history of migraines, epilepsy or traumatic brain injury.
* Have a scalp or skin condition (e.g., psoriasis or eczema), metallic implants (except for dental fillings or caps) or retained metal fragments.
* History of neurologic condition or genetic disorder associated with neurocognitive impairment unrelated to cancer diagnosis or treatment.
* Not fluent in English.
* Taking a psychoactive drug or stimulant.

Ages: 8 Years to 215 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2019-11-18 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants who completed three sessions of tDC stimulation and cognitive testing. | 12 months after participant enrollment
  The trial will be considered feasible if at least 30 survivors are able to complete 3 sessions (tDCS along with cognitive testing).

SECONDARY OUTCOMES:
Bushke selective remining test (BSRT) | 48 hours
  BSRT is a test that evaluates verbal memory performance
NIH toolbox list sorting working memory test (WM) | 48 hours
  WM is a test that evaluates information processing and storage performance
NIH toolbox flanker inhibitory control and attention test (Flanker) | 48 hours
  Flanker is a test that evaluates attention and inhibitory control
Grooved peg board test (GPB) | 48 hours
  GPB is a test that evaluates visual-motor coordination and motor speed

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas S Phillips, MD, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols